CLINICAL TRIAL: NCT05052541
Title: Safety and Efficacy of Oral Cannabis in Chronic Spine Pain
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Institute of Cannabis Research (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 20-0701
Record Dates: First submitted 2021-08-18; First posted 2021-09-22 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Back Pain; Neck Pain
MeSH Terms: conditions — Back Pain; Neck Pain | interventions — Dronabinol

STUDY DESIGN:
Intervention Model Description: One Main Arm is Crossover (Analgesia Arm) One Main Arm is Parallel (Reduction Arm)
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Analgesia Arm: THC (tetrahydrocannabinol), then THC/CBD (cannabidiol), then Placebo (Experimental): Subjects in this crossover arm will be assigned to 6 weeks on THC oral solution, then 6 weeks on THC/CBD oral solution, then 6 weeks on Placebo oral solution. Frequency of drug administration is 3-4 times a day.
  Interventions: Drug: THC/CBD; Drug: THC; Drug: Placebo
- Analgesia Arm: THC, then Placebo, then THC/CBD (Experimental): Subjects in this crossover arm will be assigned to 6 weeks on THC oral solution, then 6 weeks on Placebo oral solution, then 6 weeks on THC/CBD oral solution. Frequency of drug administration is 3-4 times a day.
  Interventions: Drug: THC/CBD; Drug: THC; Drug: Placebo
- Analgesia Arm: THC/CBD, then THC, then Placebo (Experimental): Subjects in this crossover arm will be assigned to 6 weeks on THC/CBD oral solution, then 6 weeks on THC oral solution, then 6 weeks on Placebo oral solution. Frequency of drug administration is 3-4 times a day.
  Interventions: Drug: THC/CBD; Drug: THC; Drug: Placebo
- Analgesia Arm: THC/CBD, then Placebo, then THC (Experimental): Subjects in this crossover arm will be assigned to 6 weeks on THC/CBD oral solution, then 6 weeks on Placebo oral solution, then 6 weeks on THC oral solution. Frequency of drug administration is 3-4 times a day.
  Interventions: Drug: THC/CBD; Drug: THC; Drug: Placebo
- Analgesia Arm: Placebo, then THC, then THC/CBD (Experimental): Subjects in this crossover arm will be assigned to 6 weeks on Placebo oral solution, then 6 weeks on THC oral solution, then 6 weeks on THC/CBD oral solution. Frequency of drug administration is 3-4 times a day.
  Interventions: Drug: THC/CBD; Drug: THC; Drug: Placebo
- Analgesia Arm: Placebo, then THC/CBD, then THC (Experimental): Subjects in this crossover arm will be assigned to 6 weeks on Placebo oral solution, then 6 weeks on THC/CBD oral solution, then 6 weeks on THC oral solution. Frequency of drug administration is 3-4 times a day.
  Interventions: Drug: THC/CBD; Drug: THC; Drug: Placebo
- Reduction Arm: THC/CBD (Experimental): Subjects in this parallel arm will be assigned to 13 weeks on THC/CBD oral solution. Frequency of drug administration is 3-4 times a day.
  Interventions: Drug: THC/CBD
- Reduction Arm: Placebo (Placebo Comparator): Subjects in this parallel arm will be assigned to 13 weeks on Placebo oral solution. Frequency of drug administration is 3-4 times a day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: THC/CBD — Oral solution containing 5mg THC and 50 mg CBD per 1 ml
  Arms: Analgesia Arm: Placebo, then THC, then THC/CBD; Analgesia Arm: Placebo, then THC/CBD, then THC; Analgesia Arm: THC (tetrahydrocannabinol), then THC/CBD (cannabidiol), then Placebo; Analgesia Arm: THC, then Placebo, then THC/CBD; Analgesia Arm: THC/CBD, then Placebo, then THC; Analgesia Arm: THC/CBD, then THC, then Placebo; Reduction Arm: THC/CBD
Drug: THC — Oral solution containing 5mg THC per 1 ml
  Arms: Analgesia Arm: Placebo, then THC, then THC/CBD; Analgesia Arm: Placebo, then THC/CBD, then THC; Analgesia Arm: THC (tetrahydrocannabinol), then THC/CBD (cannabidiol), then Placebo; Analgesia Arm: THC, then Placebo, then THC/CBD; Analgesia Arm: THC/CBD, then Placebo, then THC; Analgesia Arm: THC/CBD, then THC, then Placebo
Drug: Placebo — Oral solution containing no active drug
  Arms: Analgesia Arm: Placebo, then THC, then THC/CBD; Analgesia Arm: Placebo, then THC/CBD, then THC; Analgesia Arm: THC (tetrahydrocannabinol), then THC/CBD (cannabidiol), then Placebo; Analgesia Arm: THC, then Placebo, then THC/CBD; Analgesia Arm: THC/CBD, then Placebo, then THC; Analgesia Arm: THC/CBD, then THC, then Placebo; Reduction Arm: Placebo

SUMMARY:
The overall objectives of this study are to investigate the efficacy of extended cannabis treatment to reduce patient exposure to prescription opioids through its use 1) as a non-opioid analgesic treatment, and 2) as a therapy for reducing high-dose opioid use in patients with chronic spine pain.

DETAILED DESCRIPTION:
This randomized, placebo-controlled clinical trial is designed to elucidate the role of extended oral cannabis treatment in the alleviation of chronic spine pain and reduction of high-dose opioid use. This trial includes two study arms: Analgesia Arm and Reduction Arm. The Analgesia Arm uses a within-subject crossover design to determine whether daily treatment with an oral cannabis solution for 6 weeks significantly reduces spine pain compared to placebo. The Reduction Arm uses a parallel design to determine whether daily treatment with an oral cannabis solution for 13 weeks results in a greater reduction of pain and opioid intake than placebo treatment. It will also assess the impact of extended cannabis treatment on opioid craving and symptoms of opioid withdrawal in participants tapering their high-dose opioids.

ELIGIBILITY:
Some inclusion/exclusion criteria are purposely omitted at this time to preserve scientific integrity. They will be included after the trial is complete.

Inclusion Criteria:

Self-reported chronic (≥3 months' duration), non-radicular spine pain

Exclusion Criteria:

Unwilling/unable to refrain from cannabis use (medical or recreational) for 14 days prior to Baseline Visit and throughout the study (other than study drug). This includes whole plant inhalation, edibles, extracts, and topicals.

Co-morbid cancer-related pain condition

Neuropathic Pain

A co-morbid pain condition that is of greater severity than the patient's spine pain

Spine or other major surgery within the 3 months prior to enrollment

Planned surgery or procedural intervention during the study period

Allergy or adverse reaction to cannabis

Current or historical substance use disorder

Current or historical alcohol use disorder

Current or prior cannabis abuse/dependence

Positive result for use of amphetamine/methamphetamine, barbiturates, benzodiazepines, cocaine, phencyclidine (PCP), ecstasy (MDMA), as detected on urine screen

Current use of valproate, clobazam, clopidogrel, warfarin, barbiturates, benzodiazepines

Prior adverse reaction to cannabis exposure (paranoia, anxiety, etc.)

History or diagnosis of schizophrenia, bipolar or a psychotic disorder

History of any mental health illness that in the opinion of the Investigator would compromise the safety of the participant

Current or historical severe depression

Current suicidal ideation

Diagnosed cognitive impairment (e.g. Alzheimer's Disease, traumatic brain injury)

Uncontrolled hypertension (>139/89)

Abnormal values on CBC (complete blood count) or CMP (comprehensive metabolic panel) laboratory analysis that are deemed clinically significant by study physician

Known hepatic disease or dysfunction, or identification of such on screening laboratory studies

Known cardiovascular disease

Abnormal result on electrocardiogram (ECG) that is deemed clinically significant by study MD

Cognitive disability that interferes with ability to provide consent or understand study procedure

History of seizure disorder

Any medical condition for which immunosuppressive therapy is required.

Inability to refrain from using tobacco for at least 4 hours

Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the participant or the quality of the data

Pending legal action or workers compensation

Pregnant females or females intending to become pregnant during the study period

Unwilling to use one of the accepted forms of contraception during the study period and for at least 60 days after completion of the study (females of childbearing potential and males with sexual partners of childbearing potential)

Lactating females

Analgesia Arm Exclusion Criteria:

Unwilling/unable to discontinue current opioid use for 14 days prior to Baseline study visit and throughout the study

Reduction Arm Exclusion Criteria:

Not interested in reducing or discontinuing use of prescribed opioids for chronic pain

Unwilling to allow the study team to communicate with the participant's opioid prescribing provider

*Some inclusion/exclusion criteria are purposely omitted at this time to preserve scientific integrity. They will be included after the trial is complete.

Ages: 21 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change in chronic pain as measured by the Visual Analog Scale (VAS) for pain | Weekly, up to week 22
  The Visual Analog Scale (VAS) for pain is a 0-100mm visual scale anchored by "no pain" and "worst possible pain".
Change in opioid dose as measured in morphine milligram equivalents (MME) | Weekly, up to week 22

SECONDARY OUTCOMES:
Study Drug Tolerability as measured by study drug use | Daily, up to week 22
  study drug dose, frequency
Study Drug Tolerability as measured by side effects | Daily, up to week 22
Change in spine-related disability and quality of life as measured on the NIH Patient Reported Outcomes Measurement System (PROMIS)-29 | Weekly, up to week 22
  The NIH Patient Reported Outcomes Measurement System (PROMIS)-29 is a collection of 4-item short forms assessing anxiety, depression, fatigue, pain interference, physical function, sleep disturbance, and ability to participate in social roles and activities as well as a single pain intensity item.
Change in spine-related disability and quality of life as measured on the NIH Task Force on Research Standards for Chronic Low-Back/Neck Pain Minimal Dataset | Weekly, up to week 22
  The NIH Task Force on Research Standards for Chronic Low-Back Pain Minimal Dataset (and the modified Dataset for neck pain) assesses the influence of back/neck pain on physical function, emotional health, sleep, everyday activities.
Change in use of opioid and non-opioid analgesic medications | Daily, up to week 22
Change in abuse liability of cannabis as measured on the Drug Effects Questionnaire (DEQ) for study drug (cannabis) | Weekly, up to week 22
  The Drug Effects Questionnaire (DEQ) for study drug (cannabis) assesses the subjective effects after taking a drugs, including feeling a drug effect, liking/disliking the drug effect, feeling high, and wanting more drug.
Change in abuse liability of cannabis as measured on a VAS for study drug (cannabis) craving | Weekly, up to week 22
  The VAS for study drug (cannabis) craving is a 100 mm visual scale anchored by "not at all" and "extremely" when asked about drug craving in the past week
Change in opioid craving and withdrawal as measured on a VAS for opioid craving | Weekly, up to week 22
  The VAS for opioid craving is a 100 mm visual scale anchored by "not at all" and "extremely" when asked about opioid craving in the past week.
Change in opioid craving and withdrawal as measured on the Subjective Opiate Withdrawal Scale (SOWS) | Weekly, up to week 22
  The Subjective Opiate Withdrawal Scale (SOWS) is a self-report questionnaire containing 16 symptoms related to opioid withdrawal.
Change in opioid craving and withdrawal as measured on the Drug Effect Questionnaire (DEQ) | Weekly, up to week 22
  The Drug Effects Questionnaire (DEQ) for opioids assesses the subjective effects after taking opioids, including feeling a drug effect, liking/disliking the drug effect, feeling high, and wanting more opioids.
Change in opioid craving and withdrawal as measured on the Current Opioid Misuse Measure (COMM). | Weekly, up to week 22
  Current Opioid Misuse Measure (COMM) is a brief patient self-assessment to help identify participants who exhibit aberrant behaviors associated with the misuse of opioid medications.
Change in pain sensitivity as measured by pain threshold (kPa) to a pressure stimulus | Weekly, up to week 22
  Pressure output on a computer-controlled pressure algometer will be set to 10 kPa/s and participants will be instructed to indicate when the sensation changes from one of pressure alone to one of pressure and pain (pain threshold) by pressing a button on the remote-control indicator
Change in cognition as assessed by the List Sorting Working Memory Test | Weeks 5, 13 and 21 (Analgesia Arm) Week 12 (Reduction Arm)
  The List Sorting Working Memory Test measures attention/working memory. Participants recall and sequence different visually and orally presented stimuli (e.g., participants are asked to list a set of given animals in order by size, from smallest to largest).
Change in cognition as assessed by the Pattern Comparison Processing Speed Test | Weeks 5, 13 and 21 (Analgesia Arm) Week 12 (Reduction Arm)
  The Pattern Comparison Processing Speed Test is a measure of processing speed. Participants discern whether two side-by-side pictures are the same or not, with 85 seconds to respond to as many items as possible.
Change in cognition as assessed by the Oral Symbol Digit Test | Weeks 5, 13 and 21 (Analgesia Arm) Week 12 (Reduction Arm)
  The Oral Symbol Digit Test is a measure of processing speed. Symbols on the screen are associated with a number in a key. Participants are then presented symbols without numbers. Participants say each number that goes with each presented symbol for 90 seconds.
Change in cognition as assessed by the Flanker Inhibitory Control and Attention Test | Weeks 5, 13 and 21 (Analgesia Arm) Week 12 (Reduction Arm)
  The Flanker Inhibitory Control and Attention Test measures attention and inhibitory control. Participants are required to indicate the left-right orientation of a centrally presented stimulus while inhibiting attention to the potentially incongruent stimuli that surround it (i.e., the flankers, two on either side).
Change in cognition as assessed by the Picture Vocabulary Test | Weeks 5, 13 and 21 (Analgesia Arm) Week 12 (Reduction Arm)
  The Picture Vocabulary Test measures receptive vocabulary. Respondents select pictures (from arrays) that most closely match the meanings of presented words.
Change in cognition and motor skills as assessed by the Hopkins Verbal Learning Test Revised (HVLT-R) | Weeks 5, 13 and 21 (Analgesia Arm) Week 12 (Reduction Arm)
  The HVLT-R is a measure of verbal learning and memory. Participants are asked to learn a 12-item word list over three trials (total immediate learning). A delayed free recall trial is administered after 20 minutes, followed by a yes/no recognition trial.
Change in motor skills as assessed by the Grooved Pegboard Test | Weeks 5, 13 and 21 (Analgesia Arm) Week 12 (Reduction Arm)
  The Grooved Pegboard is a test of fine motor coordination and speed. In this test, participants place 25 small metal pegs into holes on a 3"x3" metal board as quickly as possible. All pegs are alike and have a ridge on 1 side that corresponds to a randomly oriented notch in each hole on the metal board.
Change in motor skills as assessed by the Standardized Field Sobriety Test | Weeks 5, 13 and 21 (Analgesia Arm) Week 12 (Reduction Arm)
  The Standardized Field Sobriety Test is intended to detect driving impairments due to recent alcohol or drug use.
Change in participant's perceived improvement in spine pain as measured on the Patient Global Impression of Change Scale (PGIC) | Weeks 5, 13 and 21 (Analgesia Arm) Week 12 (Reduction Arm)
  The Patient Global Impression of Change Scale (PGIC) is a 7-point scale depicting a patient's rating of overall improvement.

OTHER OUTCOMES:
Change in 2-arachidonoylglycerol levels as measured in plasma | Baseline, Weeks 5, 13 and 21 (Analgesia Arm) Week 12 (Reduction Arm)
  2-arachidonoylglycerol will be measured in pmol/ml
Change in N-arachidonoylethanolamine levels as measured in plasma | Baseline, Weeks 5, 13 and 21 (Analgesia Arm) Week 12 (Reduction Arm)
  N-arachidonoylethanolamine will be measured in pmol/ml
Change in tumor necrosis factor alpha (TNF-α) levels as measured in plasma | Baseline, Weeks 5, 13 and 21 (Analgesia Arm) Week 12 (Reduction Arm)
  TNF-α will be measured in pg/ml
Change in C-reactive protein (CRP) levels as measured in plasma | Baseline, Weeks 5, 13 and 21 (Analgesia Arm) Week 12 (Reduction Arm)
  CRP will be measured in mg/L

CONTACTS AND LOCATIONS:
Overall Officials: Emily Lindley, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States